CLINICAL TRIAL: NCT01536639
Title: Physiological Concept of Insulin Therapy in Subjects With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1929
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administered by subcutaneous injection. The physician determined the starting dose and frequency, as well as later changes to either dose or frequency, if any

SUMMARY:
This study is conducted in Europe. The aim of the study was to evaluate the safety and efficacy of biphasic insulin aspart 30 (NovoMix® 30) when switching to a modern premix insulin analogue treatment compared to previous insulin regimen in routine clinical practice in the Slovak Republic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with type 2 diabetes in whom at the discretion of the investigator it was decided to change insulin regimen to biphasic insulin aspart 30
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Fasting plasma glucose (FPG)
Post-prandial glucose (PPG)
Weight
Hypoglycaemia
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- [Result] Significant reduction in proportion of T2 diabetes patients at high risk for developing late complications after switching human insulin to BIAsp 30; results of an observational study in Slovakia; Z. Schroner; 2085-PO; 69th American Diabetes Association, New Orleans 2009
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com